CLINICAL TRIAL: NCT04581564
Title: Investigating the Neural Mechanisms Underlying Language Recovery Through Rhythm Therapy
Brief Title: Rhythm-based Intervention in Aphasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspension of IRB (Institutional Review Board) Approval
Sponsor: The University of Texas at Dallas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-4; R21DC018699 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-10-09 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia | interventions — Singing

STUDY DESIGN:
Intervention Model Description: The intervention is administered using an app installed in a smart phone or tablet personal computer. It does not involve drug, etc.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rhythm intervention (Experimental): Practice speech production daily through rhythmic activity
  Interventions: Behavioral: Rhythm-based speech therapy app (i.e., Speech Hero)
- Non-rhythm intervention (Active Comparator): Conventional speech production therapy without the use of rhythmic activities
  Interventions: Behavioral: Non-rhythm based (singing) application (conventional speech therapy)

INTERVENTIONS:
Behavioral: Rhythm-based speech therapy app (i.e., Speech Hero) — Participants will be issued a tablet device pre-installed with a rhythm-based application. They will initially be given a tutorial on how to use the application and encouraged to use application on a daily basis but at the least 5 times a week.
  Arms: Rhythm intervention
Behavioral: Non-rhythm based (singing) application (conventional speech therapy) — Participants will be issued a tablet device pre-installed with a singing-based application. They will initially be given a tutorial on how to use the application and encouraged to use application on a daily basis but at the least 5 times a week.
  Arms: Non-rhythm intervention

SUMMARY:
Every year, approximately 100,000 people are diagnosed with aphasia-a language disorder leading to substantial difficulties in their daily communication. Based on the observation that many people with aphasia can sing words that they otherwise cannot speak, melodic intonation therapy (MIT) was developed in the 1970s. Although recognized as a standard aphasia treatment, the neural mechanisms of MIT have been largely unexplored.

Our first goal is to identify the active ingredient of the music intervention. Although rhythm has long been considered secondary to melody, recent evidence has challenged this notion by demonstrating that rhythm alone is sufficient enough to facilitate improvements in speech fluency for people with aphasia. To corroborate the positive role of rhythm, we will train aphasic patients to leverage "rhythmic groove" for sets of sentences/phrases delivered through a fun and engaging video gaming platform. This intervention emerges from the theoretical framework, built from neuroimaging data, that language processes heavily rely on neural resources within the sensorimotor and fronto-striatal circuits that subserve rhythm/timing processes.

Our second goal is to characterize the neural plasticity associated with language recovery promoted by the novel rhythm-based therapy. We hypothesize that neuroplasticity will manifest itself as increased white matter tracts, presumably due to changes in myelination in either ipsilateral or contralateral (homologues) language areas. To effectively measure myelin white matter fraction (MWF) in candidate tracts, we will mainly use a patented Laplace-transformed relaxation MRI technique. Additionally, we will measure resting-state functional connectivity using BOLD (Blood Oxygen-Level Dependent) fMRI (functional Magnetic Resonance Imaging). Lastly, we will attempt to record cortical activity using fNIRS (functional Near-Infrared Spectroscopy) during the pre-post behavioral assessments.

Taken together, the proposed interdisciplinary research has theoretical, methodological, and clinical innovations and significance. This exploratory work will serve as a critical stepping stone toward unraveling the therapeutic component of music in neurological disorders and will provide evidence-based guidance to the clinicians and therapists.

DETAILED DESCRIPTION:
Every year, approximately 800,000 people have a stroke in the United States alone. Among these individuals, roughly 100,000 are diagnosed with aphasia-a disorder characterized by profound challenges in daily communication with their families and peers. Notably, many individuals with aphasia can sing despite their speech difficulties, an observation which led to the development of melodic-intonation therapy (MIT) in the 1970s. Although MIT has since been accepted as a viable aphasia therapy by the American Academy of Neurology, the underlying neurological mechanisms that enable speech recovery remain poorly understood. Here, we propose a highly interdisciplinary approach to study the neural mechanisms of language recovery in aphasia through a novel rhythm-based language intervention.

Our ultimate goal is to help clinicians and therapists optimize aphasia treatment by elucidating the neural basis underlying music-induced language recovery through multimodal neuroimaging and novel statistical analysis. In particular, we will test a hypothesis that rhythm alone is sufficient to facilitate language recovery, without melody To explore this hypothesis, we recently devised a novel framework for music-based language therapy that solely leverages rhythm to facilitate language production at the phrase or sentence level. Our therapy was used in a case study with a patient with chronic aphasia who had severely impaired speech fluency due to a large unilateral stroke in the left hemisphere. Following eight weeks of rhythm therapy, she exhibited remarkable improvement in speech production (i.e., from 1-2 spontaneous words to 16 sentences made from 42 words), and increased functional and structural connectivity within key regions of interest associated with the right sensorimotor network. While compelling, these preliminary data warrant further validation using proper active controls and a larger sample size, a goal to be achieved through the proposed research. We have since translated the rhythm therapy into a fun and engaging game termed "TheraBeat" that can be installed on a tablet Personal Computer or smart phone. In the proposed research, we will use TheraBeat as a home-based aphasia therapeutic intervention to minimize the burden of patient travel and increase accessibility to therapy. The proposed study will be accomplished by pursuing the following specific aims:. This prediction is based upon the theoretical and neuroscientific framework that demonstrates how language heavily relies on rhythm processes mediated by the bilateral sensorimotor network.

Aim 1. Determine the therapeutic role of rhythm in speech recovery for people with aphasia. Based on recent evidence garnered by our group as well as others, we expect that rhythm-based rehabilitation will enhance speech fluency in people with chronic aphasia, i.e., our target patients who are beyond six months after the onset of stroke. This hypothesis will be tested by directly comparing post-therapy outcomes of the treatment group, who will practice speech production daily through rhythmic activity, to an active control group who will receive conventional speech production therapy without the use of rhythmic activities.

Aim 2. Characterize the neural plasticity promoted by rhythm-based intervention. We hypothesize that daily participation in our new therapy program will promote neuroplasticity along the sensorimotor network, especially within the intact perilesional left or right fronto-striatal circuits that are known to play a key role in speech production and fluency. To determine structural neuroplasticity following the intervention, we will utilize patented myelin-based MRI in combination with diffusion tensor imaging (DTI). To explore functional neuroplasticity, we will use both resting-state fMRI and functional near-infrared spectroscopy (fNIRS). These structural and functional data will be analyzed via a novel statistical shape analysis that captures morphological changes, which cannot be detected by simple statistical approaches.

By using an innovative rhythm-based therapeutic intervention and cutting-edge neuroimaging techniques, we will address hitherto unknown questions regarding how and why music works as a therapeutic regimen for aphasia rehabilitation. With expertise in aphasia rehabilitation, neuroimaging, computer science, and data analytics, our interdisciplinary research team is well poised to undertake this investigation. The proposed research will serve as a critical stepping stone toward understanding the therapeutic role of music in neurological disorders. Our results will lay the foundations for future studies on music-induced language recovery.

ELIGIBILITY:
Inclusion Criteria:

* Must be over six months post-stroke
* Limb motor function, at least on the left side, should remain relatively intact
* Be able to name at least few items
* Must not suffer from any other type of neurological disease.

Exclusion Criteria:

* less than six months post-stroke
* Metal in the body
* Comorbidity with other neurological disorders (e.g., depression)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yune Lee, PhD, Principal Investigator — UT Dallas
Locations (1):
- Yune S Lee, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early, before reaching the anticipated enrollment. All 4 participants enrolled were assigned to the Rhythm Intervention group.
Groups:
- Rhythm Intervention: Practice speech production daily through rhythmic activity
  Rhythm-based speech therapy app (i.e., Speech Hero): Patients with non-fluent aphasia will practice speech production during the intervention period.
- Non-rhythm Intervention: Conventional speech production therapy without the use of rhythmic activities
  Rhythm-based speech therapy app (i.e., Speech Hero): Patients with non-fluent aphasia will practice speech production during the intervention period.
Period: Overall Study
Arm/Group | Rhythm Intervention | Non-rhythm Intervention
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early, before reaching the anticipated enrollment. All 4 participants enrolled were assigned to the Rhythm Intervention group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rhythm Intervention | Non-rhythm Intervention | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data collected was not analyzed following the IRB termination of the study.
  Participants
    Female | 1 | 0 | 1
    Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Aphasia Spoken Word Assessment
Description: Participants will be evaluated on practiced spoken words. The mean difference of practiced spoken words before and after the intervention will be calculated.
Time Frame: 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of practiced spoken words
Arm/Group | Rhythm Intervention | Non-rhythm Intervention
Number analyzed (Participants) | 4 | 0
Number of practiced spoken words | 1.5 (9.434) |

2. Primary Outcome: Western Aphasia Battery (WAB) Test
Description: Participants' language ability will be assessed with Western Aphasia Battery (WAB), whose reliability and validity have been well established. The mean difference before and after the intervention will be calculated. The Aphasia Quotient is scored on a scale of 0-100. Lower scores represent more severe aphasia and higher scores represent lesser aphasia severity.
Time Frame: 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rhythm Intervention | Non-rhythm Intervention
Number analyzed (Participants) | 4 | 0
score on a scale | 0.475 (0.629) |

ADVERSE EVENTS:
Time Frame: From enrollment to study completion (For a total of 6 months)
Description: Adverse event information was collected in a non-systemic manner.
Arm/Group | Rhythm Intervention | Non-rhythm Intervention
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

LIMITATIONS AND CAVEATS:
The procedures specified in the protocol were determined to be non-compliant by the IRB (Institutional Review Board) and the deviations may have compromised integrity of the data collected and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT04581564/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT04581564/ICF_001.pdf